CLINICAL TRIAL: NCT00512161
Title: A Retrospective Study to Determine the Frequency of Indications That Lead to the Placement of Permanent Pacemakers After Cardiac Surgery
Brief Title: Placement of Permanent Pacemaker Study
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 0701008942
Record Dates: First submitted 2007-08-03; First posted 2007-08-07 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Cardiac Surgical Procedures
Keywords: Any patient undergoing elective cardiac surgery

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the predictors for placement of permanent pacemakers soon after cardiac surgery. We will measure the following to see what influence, if any, they have on predicting the need for permanent pacemaker implantation.

1. Type of cardiac surgery
2. Gender of patient
3. Patient's age
4. Preoperative heart rhythm and rate
5. Duration on cardiopulmonary bypass
6. Immediate post cardiopulmonary bypass heart rhythm and rate.
7. All heart rhythms and rates identified in the postoperative period prior to permanent pacemaker implantation.
8. Underlying heart rhythm and rates when permanent pacemaker is placed.
9. Ejection fraction before surgery
10. Ejection fraction immediately post-cardiopulmonary bypass

DETAILED DESCRIPTION:
The purpose of this study is to determine the predictors for placement of permanent pacemakers soon after cardiac surgery. We will measure the following to see what influence, if any, they have on predicting the need for permanent pacemaker implantation. Through investigation into the co-morbidities, diagnoses, or histories associated with an endpoint permanent pacemaker placement, it is possible that we will garner a better idea of who will require PPP.

ELIGIBILITY:
Inclusion Criteria:

* All patients between the ages of 18-99 years.
* All patients undergoing cardiac surgery requiring cardiopulmonary bypass.

Exclusion Criteria:

* Patients who have permanent pacemakers in place.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiopulmonary Bypass Patients without a pacemaker already in place
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2007-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory E. Kerr, M.D., M.B.A., Principal Investigator — Weill Medical College of Cornell University; John J. Savarese, M.D., Study Chair — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No